CLINICAL TRIAL: NCT00232986
Title: A Comparison of Survey Methodologies to Elicit Information on Sexual and Reproductive Health From Adolescents in Urban India
Brief Title: A Comparison of Survey Methodologies to Elicit Sensitive Information From Adolescents in Urban India
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Hopkins Population Center's Mellon Grant (Unknown); Bill and Melinda Gates Foundation (Other); The Woodrow Wilson- Johnson & Johnson Dissertation Fellowship in Women's Health. (Unknown)
Other Study IDs: H.32.04.02.23.A2
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2005-10-05 (Estimated); Status verified 2005-10

CONDITIONS: Unmarried Male and Female Adolescents in the Age Group 15-19 Years in Pre-Identified Slums in Delhi, India

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The goal of this study is to use three different survey methodologies to evaluate whether adolescents report on their knowledge, attitudes and behaviors on sexual and reproductive health issues differently based on the manner in which questions are asked.

DETAILED DESCRIPTION:
Specific Aims and Research Questions Aim 1: To compare adolescents' levels of reporting of their own reproductive health knowledge, attitudes and behaviors using three survey methodologies: (1) Face-to-face interview (2) Audio-CASI (Computer Assisted Self Interview) and (3) a culturally appropriate interactive methodology.

The following hypothesis will be tested:

• Overall, adolescents will be more likely to divulge their own reproductive knowledge, attitudes and behaviors with Audio-CASI and the interactive method as compared to face-to-face interviews. Levels of knowledge, attitudes and behaviors will vary by education, age and gender.

Aim 2: To compare respondents' levels of comfort, accuracy and honesty with the survey methodologies (i.e. face to face, audio-CASI and interactive methodology) to their reporting of knowledge, attitudes and behaviors related to sexual and reproductive health.

ELIGIBILITY:
Inclusion Criteria:

Unmarried male and female adolescents in the age group 15-19 in pre-identified slums in Delhi, India

Exclusion Criteria:

-

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 960
Dates: Start 2004-09; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Hindin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health